CLINICAL TRIAL: NCT02937831
Title: RIXUBIS Drug Use-Result Survey (Japan)
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 251601
Record Dates: First submitted 2016-10-05; First posted 2016-10-19 (Estimated); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Study Participants
  Interventions: Biological: RIXUBIS

INTERVENTIONS:
Biological: RIXUBIS
  Other Names: Coagulation Factor IX [Recombinant]; BAX 326; Recombinant factor IX; BAX326

SUMMARY:
The purpose of this survey is to understand the following items observed in the actual clinical use of RIXUBIS.

1. Unexpected adverse drug reactions
2. Occurrence of adverse drug reactions in the actual clinical use
3. Factors that may affect safety and effectiveness
4. Occurrence of Factor IX (FIX) inhibitor development in patients with coagulation FIX deficiency
5. Safety and effectiveness for hemophilia B patients who received routine prophylactic therapy, on-demand therapy and perioperative therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia B scheduled to receive treatment with RIXUBIS

Exclusion Criteria:

* Patients not administered RIXUBIS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia B (congenital blood coagulation factor IX deficiency) who receive RIXUBIS in the actual clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (5):
- Japan (5):
  - Seki-shi, Japan, Seki-shi, Gifu
  - Maebashi-shi, Japan, Maebashi, Gunma
  - Nobeoka-shi, Japan, Nobeoka-shi, Miyazaki
  - Niigata-shi, Japan, Niigata, Niigata
  - Osaka-shi, Japan, Osaka, Osaka

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc64db2bf003ab45dff?idFilter=%5B%22251601%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 2 investigative sites in Japan, from November 16, 2016 to May 11, 2022.
Pre-assignment Details: Participants with a historical diagnosis of hemophilia B were enrolled. Participants received Nonacog Gamma (Genetical Recombination) as part of a routine medical care.
Groups:
- Nonacog Gamma (Genetical Recombination): Nonacog Gamma (Genetical Recombination) is reconstituted with the attached 5 mL reconstitution diluent and administered by intravenous injection. Do not infuse any faster than 10 mL per minute. Normally, administer 50 international units per kg body weight per time. Adjust a dose based on a participant's condition. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Nonacog Gamma (Genetical Recombination)
Started | 6
Completed | 2
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued the Use of Nonacog Gamma (Genetical Recombination)
Description: Number of participants who discontinued the use of Nonacog Gamma (Genetical Recombination) was reported in this outcome measure.
Time Frame: Throughout the study period, approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 2
Participants | 1

2. Primary Outcome: Number of Participants Who Developed a Factor IX (FIX) Inhibitor
Description: Number of participants who developed a Factor IX (FIX) Inhibitor was reported in this outcome measure.
Time Frame: Throughout the study period, approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 2
Participants | 0

3. Primary Outcome: Annual Bleed Rate (ABR): Number of Times of Bleeding During the Study
Description: Annual bleed rate (ABR) was defined as the number of times of bleeding during the study. ABR was reported in this outcome measure.
Time Frame: Throughout the study period, approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed is the number of participants who received routine prophylactic therapy.
Measure: Mean (Standard Deviation); unit: bleeds
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 1
bleeds | 0 (NA) — The standard deviation was not evaluable due to low number of participants with events.

4. Primary Outcome: Number of Doses to Treat A Bleed of Participants on An On-Demand Regimen
Description: Number of doses to treat a bleed of participants on an on-demand regimen was reported in this outcome measure.
Time Frame: At bleed resolution throughout the study period of approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed is the number of participants who received an on-demand regimen.
Measure: Number; unit: doses
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 1
doses | 1

5. Primary Outcome: Hemostatic Effectiveness of Rixubis for Participants on An On-Demand Regimen Based on a 4-Point Ordinal Scale (Excellent, Moderate, Good, Poor)
Description: Number of participants in hemostatic effectiveness of Rixubis with a 4-point ordinal scale (Excellent, Moderate, Good, Poor) for an on-demand regimen was reported in this outcome measure. The definition of each scale was following: Excellent; After a single infusion, complete disappearance of pain and objective decrease of bleeding symptom (swelling, tenderness, and increase in range of motion in musculoskeletal bleeding case) were observed. Good; After a single infusion, there were definitive relief of pain and improvement of bleeding symptom. Fair; After a single infusion, there were a probable or slight relief of pain and a mild improvement of bleeding signs. Poor; Improvement was not observed or symptom was aggravated.
Time Frame: At bleed resolution throughout the study period of approximately 4 ½ years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 1
Participants
  Excellent | 1
  Good | 0
  Moderate | 0
  None | 0

6. Primary Outcome: Hemostatic Effectiveness of Rixubis in Surgery-Perioperative and Postoperative Based on a 4-Point Ordinal Scale (Excellent, Moderate, Good, Poor) for Participants Who Received Perioperative Therapy During the Study
Description: Number of participants in hemostatic effectiveness of Rixubis with a 4-point ordinal scale (Excellent, Moderate, Good, Poor) for perioperative therapy was reported in this outcome measure. The definition of each scale was following: Excellent; Amount of bleeding is smaller than expected. Good; Amount of bleeding is within the expected range. Fair; Amount of bleeding is greater than expected, with use of additional concomitant medication. Poor; Hemostasis difficulty.
Time Frame: Assessed at the time of discharge from recovery room; and at 24 to 72 hours postoperatively
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed is the number of participants who received perioperative therapy. Number of participants who received perioperative therapy during this study was zero (N=0).
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Who Experienced Adverse Events of Shock or Anaphylaxis
Description: Number of participants who experienced adverse events of shock or anaphylaxis was reported in this outcome measure.
Time Frame: Throughout the study period, approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Number of Participants Who Experienced Adverse Events of Thromboembolism
Description: Number of participants who experienced adverse events of thromboembolism was reported in this outcome measure.
Time Frame: Throughout the study period, approximately 4 ½ years
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Nonacog Gamma (Genetical Recombination)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period, approximately 4 ½ years
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Nonacog Gamma (Genetical Recombination)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nonacog Gamma (Genetical Recombination) (N=2)
Upper respiratory tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02937831/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02937831/SAP_001.pdf